CLINICAL TRIAL: NCT04438746
Title: Alleviating Pain and Opioid Dependence Through Anger Management: A Pilot Study
Brief Title: Chronic Pain, Opioids, and Anger Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas at San Antonio (Other)
Responsible Party: Principal Investigator, Ephrem Fernandez, Professor, Psychology, The University of Texas at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #20-002
Record Dates: First submitted 2020-05-28; First posted 2020-06-19 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Anger; Opioid Use; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving CBAT (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Affective Therapy
- Group receiving general emotion training (Placebo Comparator)
  Interventions: Behavioral: Emotion discussion

INTERVENTIONS:
Behavioral: Emotion discussion — General discussion of emotions; no therapy or training is offered
  Arms: Group receiving general emotion training
Behavioral: Cognitive Behavioral Affective Therapy — Active training in regulating anger
  Arms: Group receiving CBAT

SUMMARY:
The current US opioid epidemic is a pressing public health concern. Links between opioid misuse and mortality are well-known; nearly 70% of all drug overdose deaths in 2017 were attributable to opioids. Given their pain-relieving properties, opioids have been widely used in the chronic pain population who are also susceptible to misuse of these analgesics.. In chronic pain patients with anger, the pain as well as opioid use may be aggravated. For example, suppression of anger has been linked with increased pain sensitivity in experiments, while anger-hostility scores and internalized anger predict pain severity variance and pain intensity, respectively. Anger is also linked with drug use/abuse, including opioids. The goal of this research is to implement a state-of-the-art program for anger regulation in chronic pain patients., Called Cognitive Behavioral Affective Therapy (CBAT), this program is evaluated on multiple measures of anger, sensory versus affective measures of pain, and measures of opioid misuse. CBAT is expected to reduce anger, and thereby produce reduction in pain as well as shift attitudes away from opioid misuse..

DETAILED DESCRIPTION:
Participants will be recruited by electronic announcements and IRB approved recruitment flyers in local pain clinics and pain support groups. These ads and flyers will contain relevant info (e.g., study email address and GoogleVoice number) for prospective participants to contact study staff with any questions about participation. Interested participants will be screened by an RA on the phone using the following steps: 1) RA will obtain verbal consent upon explaining study participation and answering any questions participants may have; 2) Once informed consent is obtained, RA will use participants preferred email address to send potential participant a link to the Qualtrics screening questionnaire; 3) RA will then briefly orient participant to Qualtrics; and 3) RA will complete the screening process with participant on the phone to determine and inform participant of their eligibility to participate.

Consent and Screening: Participants will first go through the informed consent procedure, where they will be told about the purpose of the study, expectations of them as participants, etc. Informed consent is expected to take no more than 5 minutes. They will then be asked to complete a screening questionnaire which is expected to take no more than 3 minutes. Eligible participants will be randomly assigned to one of two groups: 1) Control and 2) CBAT. Both control group and experimental group participants will be required to complete 2 pre-recorded sessions per week lasting 1 hour each (total of 8 hours) over the course of 4 weeks.

Online Sessions and Surveys: After questionnaires (including measures of pain and opioid use, the Anger Parameters Scale) have been administered at pre-treatment, the first session will serve as orientation to self-monitoring anger levels between sessions. If a participant has no anger on a given day, no monitoring is necessary. Following this, control group participants self-monitor their anger and watch pre-recorded sessions on emotions in general. The treatment group will be actively trained in anger regulation skills within the framework of CBAT. These participants will proceed from a week of anger prevention to a week of intervention to a week of postvention. During the prevention phase, an individually-tailored behavior contract against anger will be signed by each paParticipants will work with investigators over email to draft and electronically sign their contracts. RAs will review participant progress toward fulfillment of contracts during weekly check-in phone calls to participants. Participants will also engage in behavioral rehearsal of anger-provoking situations and learn about stimulus control for discriminating and avoiding situations that are likely to culminate in anger.

In the Intervention phase, participants will be introduced to techniques for regulating anger that could not be prevented. These include thought-stopping, distraction, and cognitive reappraisal..

In the postvention phase, participants will be trained in techniques for ameliorating residual anger. These include expressive writing and verbal disclosure. Gestalt therapy empty chair dialogue will be used for overcoming unresolved anger.

At the conclusion of the 4 weeks of anger self-regulation training, the same questionnaires relating to anger, pain, and opioid misuse and beliefs will be assessed in both groups. This post-treatment set of questionnaires is expected to take no more than 20 minutes.

Finally, a follow-up session (2 hours) will be held for both groups one month after post-treatment. Anger, pain, and opioid use measures will be re-administered (taking no more than 20 minutes). All participants will receive a brief booster session to reinforce effective anger regulation techniques. The same pre- and post-treatment questionnaires mentioned above will be re-administered at this point in the study.

Phone Calls and Knowledge Tests: To ensure that participants are paying attention to the online videos, RAs will contact them weekly and administer a brief, multiple choice knowledge test over the phone. Participants who score less than 50% in any given week will be dropped from the study. During that same phone call, RAs will check in with participants to ensure that there are no problems with their participation in the study and that the participants are not in any emotional distress. Phone calls are anticipated to last approximately 10 minutes, for a total time of 50 minutes over the span of the study (4 weeks of either treatment or control and the 1-month follow up). Total participant time commitment over the course of the study is approximately 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* taking opioid pain relievers for at least 3 months in the past 12 months
* maladaptive levels of anger as measured by STAXI-2
* without psychiatric co-morbidity (e.g., major depression, substance use disorder, etc.)
* not undergoing current psychological/psychiatric treatment
* speak English.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain medication dosage and frequency of use at one month | One month
  Participants are asked what pain medication they are using and at what dosage and frequency. Open-ended question.
Change in pain medication dosage and frequency of use at one month follow-up | One month after end of intervention
  Participants are asked what pain medication they are using and at what dosage and frequency. Open-ended question.
Change in attitudes/beliefs surrounding pain medication at one month | One month
  Assessed using the Pain Medication Beliefs Questionnaire (Schieffer et al., 2005), a five-item instrument measuring beliefs about one's response to, relief from, and potential addiction to pain medication
Change in attitudes/beliefs surrounding pain medication at one month follow-up | One month after end of intervention
  Assessed using the Pain Medication Beliefs Questionnaire (Schieffer et al., 2005), a five-item instrument measuring beliefs about one's response to, relief from, and potential addiction to pain medication
Change in opioid misuse at one month | One month
  Measured with the Current Opioid Misuse Measure (Butler et al., 2007), a 17-item instrument assessing signs and symptoms of drug misuse, emotional/psychiatric problems due to misuse, evidence of lying about drug use, and other domains
Change in opioid misuse at one month follow-up | One month after end of intervention
  Measured with the Current Opioid Misuse Measure (Butler et al., 2007), a 17-item instrument assessing signs and symptoms of drug misuse, emotional/psychiatric problems due to misuse, evidence of lying about drug use, and other domains
Change in anger parameters at one month | One month
  The Anger Parameters Scale taps into five parameters: Frequency, Duration, Intensity, Latency, and Threshold (Fernandez et al., 2014). Scores can range from 0-120 and higher scores imply more maladaptive anger.
  The APS is comprised of 30 items rated from 0-4. The total possible score ranges from 0 to 120. A higher score on the APS indicates more maladaptive anger.
Change in anger parameters at one month follow-up | One month after end of intervention
  The Anger Parameters Scale taps into five parameters: Frequency, Duration, Intensity, Latency, and Threshold (Fernandez et al., 2014). Scores can range from 0-120 and higher scores imply more maladaptive anger.
Change in anger expression style at one month | One month
  Measured with the Anger Expression Scale (Fernandez, 2008). The AES is comprised of 60 items rated from 0-4. These items are organized into 12 sub-scales of 5 items each. These sub-scales have a minimum total possible score of 0 and a maximum of 20. Higher scores on each sub-scale (as well as a higher cumulative score) indicates more maladaptive anger.
Change in anger expression style at one month follow-up | One month after end of intervention
  Measured with the Anger Expression Scale (Fernandez, 2008). The AES is comprised of 60 items rated from 0-4. These items are organized into 12 sub-scales of 5 items each. These sub-scales have a minimum total possible score of 0 and a maximum of 20. Higher scores on each sub-scale (as well as a higher cumulative score) indicates more maladaptive anger.
Change in chronic pain ratings at one month | One month
  Single item measured on a scale from 0-10
Change in chronic pain ratings at one month follow up | One month after end of intervention
  Single item measured on a scale from 0-10
Change in emotional response to chronic pain at one month | One month
  Single item measured on a scale from "a little unpleasant" to "extremely distressing"
Change in emotional response to chronic pain at one month follow-up | One month after end of intervention
  Single item measured on a scale from "a little unpleasant" to "extremely distressing"

CONTACTS AND LOCATIONS:
Overall Officials: Ephrem Fernandez, PhD, Principal Investigator — University of Texas at San Antonio
Locations (1):
- University of Texas at San Antonio, San Antonio, Texas, United States